CLINICAL TRIAL: NCT06008236
Title: The Effect of Progressive Muscle Relaxation and Deep Breathing Exercises Accompanied by Music on the Stress Levels of Nursing Students and Their Bio-psycho-social Responses to Stress
Brief Title: The Effect of Progressive Relaxation and Breathing Exercises Accompanied by Music on the Stress Levels of Nursing Students and Their Bio-psycho-social Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBU-NK-01
Record Dates: First submitted 2023-08-12; First posted 2023-08-23 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Stress; Stress, Physiological
Keywords: Progressive muscle exercises; Breathing; Stress
MeSH Terms: conditions — Respiratory Aspiration | interventions — Autogenic Training; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: A comparison of the two groups to be assigned as experimental and control groups will be made.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Researcher will be applied progressive muscle relaxation and deep breathing exercises to the students in the experimental group. This practice will be applied to students once a week for six weeks. It will be ensured that the environment is quiet, at room temperature and dim. Students will take their places in chairs at an equal distance from each other. The researcher will be located in a place where his voice is heard by all students, and computers and speakers will be used for music. In addition, black eye patches will be distributed to students to use while exercising before starting the exercises. The muscle groups that are desired to be contracted and relaxed will be as follows (hands, arms, muscles in the face, tongue, head and neck muscles, shoulders, waist, abdominal leg muscles, and feet). At the same time, Lily's Theme which was selected by using the literature and expert opinion, will be played to the students together with the exercises.
  Interventions: Behavioral: Progressive Muscle Relaxation and Breathing Exercises
- Control Group (No Intervention): No intervention will be applied to the control group. They will be expected to refill the scales at the end of six weeks and on the eighth week for follow-up purposes.

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation and Breathing Exercises — Progressive relaxation exercise is a method that provides relaxation in the whole body by voluntary, regular relaxation of large muscle groups in the human body. Exercise helps individuals to be able to feel the difference between tension in the muscles and relaxation, and to learn to relax on their own in case of tension. Deep breathing exercise supports the maximum ventilation of the lung by correct breathing using the diaphragm.
  Arms: Experimental Group

SUMMARY:
This clinical study will be conducted to determine the effects of musically accompanied progressive muscle relaxation and deep breathing exercises on nursing students' stress levels and bio-psycho-social responses to stress.

Do musical progressive muscle relaxation and deep breathing exercises have an impact on nursing students' stress levels and bio-psycho-social responses to stress?

After students fill in the scales, they will be randomly assigned to the experimental and control groups. The experimental group will be given progressive muscle relaxation and deep breathing exercises accompanied by music once a week for six weeks by the researcher. There will be no intervention in the control group. The scales will be reapplied to the experimental and control groups in the week after the application is completed and two weeks after the application is completed. Groups will be compared and statistical analyzes will be made.

DETAILED DESCRIPTION:
Stress is a psychosocial factor that affects students' academic performance and well-being. The presence and level of stress have a positive or negative impact on learning and thinking, and students show behavioral, emotional, and physical symptoms of experiencing stress For this reason, it is very important for university students to apply stress reduction methods, especially non-drug methods. Progressive relaxation and deep breathing exercises with music are effective methods of coping with stress. When the literature is examined, it is seen that the use of music has recently been effective in reducing the anxiety and stress experienced by many students during the education process. At the same time, a progressive relaxation exercise integrated with deep breathing exercises helps a person to feel the difference between tension and laxity in the body and allows the person to learn to relax on their own, thus reducing physical and emotional tension. Thus, the individual moves away from disturbing stimuli that reduce the quality of life such as anxiety, pain, and stress. In accordance with the nursing education program carried out with theoretical and practical application course hours, students considering the stress they are exposed to and the behavioral, emotional, and physical problems that arise with stress, there is a need for research that uses mind-body applications to support nursing students. At the end of the research, it is foreseen that the stress levels of nursing students and the symptoms seen due to stress can be reduced.

Method: The universe of the study will consist of 2nd, 3rd, and 4th year nursing undergraduate students who are studying and interning at Gülhane Nursing Faculty of Health Sciences University in 2022-2023. As a result of the power analysis, the minimum sample size was found to be 140 students, with 70 students in each group. During the study, in order to strengthen the results of the research and increase reliability, it was determined that the sample was 154 students with 77 experiments and 77 control groups with an increase of at least 10%. Student sampling; After each class is evaluated as a layer, proportional stratification will be taken by sampling method according to layer weight (number of students). 44 students from 2nd grade, 52 students from 3rd grade, and 58 students from 4th grade will participate in the research. Students have completed the Voluntary Consent Form for Nursing Students, Personal Information Form, Perceived Stress, and Bio-psycho-social Response Scale, then students who meet the inclusion criteria will be randomly assigned to intervention and control groups. Exercises will be applied to the intervention groups for 6 weeks. There will be no intervention in the control group. At the end of 6 weeks and 2 weeks after the last application (8. Weeks) intervention and control groups will refill the scales.

ELIGIBILITY:
Inclusion Criteria:

* To be a nursing student who is studying at Gulhane Nursing Faculty of Health Sciences University and going on internship
* Not to have any obstacles in oral and written communication in Turkish
* Volunteering to participate in research

Exclusion Criteria:

* If the student has a disease that prevents the relaxation exercise (Heart Failure, Musculoskeletal System Problem, etc.)
* The student is participating in another relaxation program
* The student is taking a psychiatric medication that has a relaxing effect

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | Scale; It is applied to all groups before the application starts, in the week when the application is completed (sixth week) and two weeks after the application is completed (eighth week).
  The Perceived Stress Scale for Nursing Students scale is used to determine the level of stress that nursing students perceive in their clinical practice experiences.

SECONDARY OUTCOMES:
Bio-psycho-social Response | Scale; It is applied to all groups before the application starts, in the week when the application is completed (sixth week) and two weeks after the application is completed (eighth week).
  The Bio-psycho-Social Response Scale for Nursing Students is used to determine the bio-psycho-social responses of nursing students to stress.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Yüksel, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No